CLINICAL TRIAL: NCT03239067
Title: Comparison of Short- and Long-term Efficacy and Safety Between Ticagrelor and Clopidogrel in Chinese Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention
Brief Title: Comparison Of Efficacy and Safety Between Ticagrelor and Clopidogrel In Chinese
Acronym: COSTIC
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Prof., Tongji Hospital
Other Study IDs: TJH-COSTIC
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Ticagrelor; Clopidogrel; Acute Coronary Syndrome; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

GROUPS / COHORTS (2):
- ticagrelor group: patients prescribed with ticagrelor
- clopidogrel group: patients prescribed with clopidogrel

SUMMARY:
This is a prospective, single-center study to assess the long- and short-term outcomes of ticagrelor vs clopidogrel in Chinese patients with acute coronary syndrome undergoing percutaneous coronary intervention. Patients will undergo face-to-face interviews, phone calls, or/and chart reviews at 7 days, 1 month, 6 months and 12 months. When 4500 patients have completed the follow-up, an interim analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. diagnosed as acute coronary syndrome;
3. underwent successful percutaneous coronary intervention.

Exclusion Criteria:

1. participate in any drug clinical trials within 3 months;
2. patients with life-threatening complications, or the researchers determined that the survival time of patients with no more than 1 years;
3. serious neurological disease (Alzheimer's disease, Parkinson syndrome, progressive lower limbs or deaf patients);
4. previous history of cancer or tumor, or pathological examination confirmed precancerous lesions (such as breast ductal carcinoma in situ, or atypical hyperplasia of the cervix);
5. patients refused to comply with the requirements of this study to complete the research work.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with acute coronary syndrome undergoing percutaneous coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 9040 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2021-10-24 (Actual)

PRIMARY OUTCOMES:
Composite incidence of vascular death, myocardial infarction and stroke | up to 12 months
  1. Vascular death was defined as death from cardiovascular causes or cerebrovascular causes and any unknown death unless there was another certain cause.
  2. The definition of myocardial infarction was consistent with the Third Universal Definition of Myocardial Infarction (1).
  3. Stroke was defined as a rapid onset of a new focal loss of neurologic function caused by an ischemic central nervous system event with residual symptoms lasting at least 24 hours from their onset or leading to death.

SECONDARY OUTCOMES:
Composite incidence of all-cause death, myocardial infarction and stroke | up to 12 months
  1. All-cause death was defined as any death at hospital or after discharge.
  2. The definition of myocardial infarction was consistent with the Third Universal Definition of Myocardial Infarction.
  3. Stroke was defined as a rapid onset of a new focal loss of neurologic function caused by an ischemic central nervous system event with residual symptoms lasting at least 24 hours from their onset or leading to death.
Composite incidence of vascular death, myocardial infarction, stroke, recurrent ischemia, transient ischemic attack, or other arterial thrombotic events | up to 12 months
  1. Vascular death was defined as death from cardiovascular causes or cerebrovascular causes and any unknown death unless there was another certain cause.
  2. The definition of myocardial infarction was consistent with the Third Universal Definition of Myocardial Infarction (1).
  3. Stroke was defined as a rapid onset of a new focal loss of neurologic function caused by an ischemic central nervous system event with residual symptoms lasting at least 24 hours from their onset or leading to death.

OTHER OUTCOMES:
Incidence of safety endpoints | up to 12 months
  Safety endpoints were defined according to the TIMI bleeding criteria.(2) Major bleeding (not related to heart surgery) was defined as fatal-, or intracranial bleeding including any clinically overt signs of hemorrhage associated with a decreased hemoglobin levels (≥5g/dl). Minor bleeding was defined as any clinically overt bleeding leading to decrease in hemoglobin levels of 3 to 5 g/dL or any bleeding requiring medical intervention. Minimal bleeding was defined as any overt bleeding event that did not meet the above criteria. An independent blinded central committee adjudicated all suspected endpoint event.

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, Doctor, Study Chair — Tongji Hospital,Wuhan, Hubei, China, 430030
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Derived] Hu S, Yan H, Sun Y, Wang D, Zeng H, Cui G. Triglyceride glucose index in patients with acute coronary syndrome undergoing percutaneous coronary intervention predicts cardiovascular events: a cohort study. Cardiovasc Diabetol. 2025 Oct 1;24(1):380. doi: 10.1186/s12933-025-02937-9. PMID 41034995
- [Derived] Sun Y, Li C, Zhang L, Yu T, Ye H, Yu B, Tao M, Jiang J, Yan J, Wang Y, Zeng H, Shen X, Wang DW. Clinical outcomes after ticagrelor and clopidogrel in Chinese post-stented patients. Atherosclerosis. 2019 Nov;290:52-58. doi: 10.1016/j.atherosclerosis.2019.09.011. Epub 2019 Sep 21. PMID 31568962